CLINICAL TRIAL: NCT03970434
Title: Clinical Trial to Evaluate Drug Concentration of Metformin According to Sampling Method in Healthy Adult Volunteers
Brief Title: Drug Concentration of Metformin According to Sampling Method
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Min-Gul Kim, MD, PhD, Center for Clinical Pharmacology, Chonbuk National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUH_2019_MSM
Record Dates: First submitted 2019-05-17; First posted 2019-05-31 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental)
  Interventions: Other: Venous blood collection; Other: Peripheral blood collection

INTERVENTIONS:
Other: Venous blood collection — Venous blood collection
Other: Peripheral blood collection — Peripheral blood collection

SUMMARY:
This study assess the drug concentration of metformin in healthy adult volunteers according to the sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who, at the time of screening, are the age of older than 19 years
* Subjects who have BMI more than 17.5kg/m2 and less than 30.5kg/m2 and body weight more than 55kg
* There is no congenital disease or within 3 years of chronic diseases
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, ECG or clinical laboratory tests
* Subjects who signed and dated the informed consent form(approved by IRB) after understanding fully to hear a detailed explanation in the clinical trial

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* A subject with any history of gastrointestinal disease (e.g., Crohn's disease, acute or chronic pancreatitis, and others) and surgery (except for simple appendectomy or repair of a hernia), which can influence the absorption of investigational products
* A subject who has the following clinical laboratory test results Liver Function Test (AST, ALT) > two times the upper limit of the normal range
* History of regular alcohol consumption exceeding 210g/week(12g = 125 mL of wine, 10g = 250 mL of beer, 10g = 50 mL of hard liquor) within 6 months of Screening
* A subject who has participated in any other clinical trials and had medication within 3 months prior to the first administration of investigational product.
* A subject with a history of drug abuse or a positive urine drug screening for drug abuse within 1 year
* A subject who has taken the drugs that induce and suppress drug- metabolizing enzymes within 30 days prior to investigational product administration
* A smoker who consumes more than 20 cigarettes/day within 6 months
* A subject who has taken any ethical-the-counter drug or has taken any over- the-counter drug within 10 days before the investigational product administration
* A subject who has donated whole blood within 2 months or blood components within 1 month prior to the investigational product administration
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Concentration of Metformin | 10 hours
  Compare the concentration of Metformin measured from Venous blood collection and Peripheral blood collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea